CLINICAL TRIAL: NCT01015859
Title: A Prospective Canadian Multi-center Randomized Study of the Benefits of Spontaneous Atrioventricular Conduction (Can Save R)
Brief Title: Spontaneous Atrioventricular Conduction Preservation
Acronym: CAN-SAVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Sorin Group Canada (Industry)
Responsible Party: Principal Investigator, Bernard Thibault, Cardiologist, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol IGxD04
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Patients With Pacemaker With Conduction Problems
Keywords: AV conduction; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DDD long AV delay (No Intervention): Pacemaker is programmed in DDD mode with long AV delay (250 msec)
- AAI SafeR (Active Comparator): Pacemaker is programmed in AAI SafeR mode
  Interventions: Device: Pacing mode

INTERVENTIONS:
Device: Pacing mode — To determine which mode (DDD vs AAI SafeR)minimizes ventricular pacing
  Arms: AAI SafeR

SUMMARY:
The aims of this study are to assess the clinical benefits resulting from SafeR by comparison with standard dual chamber programming (DDD) with a long atrioventricular (AV) delay.

The benefits will be assessed by comparing the percentage of ventricular pacing, the incidence of atrial arrhythmias, and the evolution of the hemodynamic status as observed through echo parameter and atrial natriuretic peptide/brain natriuretic peptide (ANP/BNP) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who fulfils one or more of the official guidelines to be implanted with a dual-chamber pacemaker (primo-implantation3) may be included in the study.

Exclusion Criteria:

The patients presenting with one or more of the following characteristics cannot be included:

Permanent complete AV block

* Permanent atrial and/or ventricular arrhythmias
* already implanted with a cardioverter-defibrillator (ICD)
* Likely to have a cardiac surgery in the next six months, mainly for:
* severe coronary artery disease
* severe valvular disease
* AV node ablation
* Refuses to sign an consent form after having received the appropriate information
* Refuses to co-operate
* Not able to understand the study objectives and protocol
* Not available for scheduled follow-up
* With a life expectancy less than one year
* Already included into another clinical study competing with the objectives of the CAN-SAVE R study
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2006-06; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
to evaluate the effectiveness of SafeR | 1 and 3 years
preserve natural AV conduction compared to DDD Long AVD | 1 and 3 years
demonstrate the effectiveness of SafeR to reduce AF incidence on a LT basis | 1 and 3 years
compare the effects of SafeR vs DDD Long AVD on LV function | 1 and 3 years

SECONDARY OUTCOMES:
total mortality | 1 and 3 years
CHF-related mortality & hospitalisations | 1 and 3 years
evolution of systemic BP | 1 and 3 years
AF-related AEs | 1 and 3 years
evolution of cardiac asynchrony [interventricular (RV-LV) & intraventricular (4 segments) | 1 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Thibault, MD, Principal Investigator — Montreal Heart Institute, Research Centre
Locations (9):
- Canada (9):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Edmonton, Alberta
  - Kingston Hospital, Queens University, Kingston, Ontario
  - Southlake Regional Hospital, Newmarket, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie, Québec, Quebec
  - Hôtel-Dieu de St Jérome, Saint Jérome, Quebec
  - Centre hospitalier régional de Trois-Rivières, Trois-Rivières, Quebec
  - Royal University Hospital, Saskatoon, Saskatoon, Saskatchewan